CLINICAL TRIAL: NCT02318394
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Clinical Activity of MEDI0562 in Adult Subjects With Selected Advanced Solid Tumors
Brief Title: A Phase 1 Study of MEDI0562 in Adult Subjects With Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6060C00001
Record Dates: First submitted 2014-12-03; First posted 2014-12-17 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; immunotherapy; OX40; immuno-oncology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monotherapy Arm (Experimental): MEDI0562 monotherapy
  Interventions: Biological: MEDI0562

INTERVENTIONS:
Biological: MEDI0562 — Subjects will receive MEDI0562 until unacceptable toxicity, confirmed disease progression or other reason for treatment discontinuation develops.

SUMMARY:
To evaluate the safety and tolerability of MEDI0562 in adult subjects with selected advanced solid tumors

DETAILED DESCRIPTION:
This is a first-time-in-human (FTiH) Phase 1, multicenter, open-label, dose-escalation, and dose-expansion study of MEDI0562 to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, pharmacodynamics and preliminary anti-tumor activity in adult subjects with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have confirmed advanced solid tumor and have progressed, are refractory, or are intolerant to standard therapy appropriate for tumor type. Subjects should not have received more than 3 prior lines of therapy for recurrent or metastatic disease including both standards of care and investigational therapies.
* Subjects must have at least 1 measurable lesion.
* Consent to provide archived tumor specimens
* Willingness to undergo pre-treatment and on-treatment biopsy.
* Adequate organ function.
* Use of highly effective contraception (females) or male condom plus spermicide (males).

Exclusion Criteria:

* Prior treatment with TNFRSF agonists.
* Subjects who have received certain prior immunotherapy or had toxicities relating to prior immunotherapy may not be permitted to enroll.

  o Must not have required the use of additional immunosuppression other than corticosteroids for the management of an adverse event.
* History of severe allergic reactions to any unknown allergens or any components of the study drug formulations.
* Receipt of any conventional or investigational anticancer therapy within 28 days prior to the first dose of MEDI0562.
* Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment.
* Unresolved toxicities from prior anticancer therapy.
* Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | From time of informed consent through 12 weeks after last dose of MEDI0562
  The maximum tolerated dose/maximum administered dose will be determined by the number of participants experiencing DLTs. The safety profile will be assessed through number of participants experiencing AEs, SAEs, abnormal laboratory parameters, vital signs and electrocardiogram (ECG) results.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated to be from time of informed consent up to 5 years
  The ORR is defined as the proportion of subjects with confirmed immune related (ir)CR or confirmed irPR
Maximum observed concentration (Cmax), area under the curve (AUC), clearance (CL) and terminal half-life of MEDI0562 | From first dose of MEDI0562 through to 30 days after last dose of investigational product
  The endpoints for assessment of PK of MEDI0562 include MEDI0562 concentrations in serum at different timepoints after MEDI0562 administration.
Number and percentage of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of MEDI0562 through to 30 days after last dose of investigational product
  The immunogenicity of MEDI0562 will be assessed by summarizing the number and percentage of subjects who develop detectable anti-drug antibodies (ADAs)
Induction of proliferation markers on various lymphocyte subsets, immunohistochemistry of tumor biopsies and assessment of programmed death ligand 1 (PD-L1) and tumor-infiltrating lymphocyte phenotypic markers | From time of informed consent through 12 weeks after last dose of investigational product
  The endpoints for assessment of pharmacodynamic activity include induction of proliferation markers in various lymphoctye subsets, immunohistochemistry of tumor biopsies and assessment of programmed death ligand 1 (PD-L1) and tumor-infiltrating lymphocyte phenotypic markers
Disease control rate (DCR) | Estimated to be from time of informed consent up to 5 years
  The DCR is defined as the proportion of subjects with irCR, irPR, or irSD (subjects achieving irSD will be included in the DCR if they maintain irSD for ≥8 weeks)
Duration of response (DoR) | Estimated to be from time of informed consent up to 5 years
  Duration of response will be defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Estimated to be from time of informed consent up to 5 years
  Progression-free survival will be measured from the start of treatment with MEDI0562 until the first documentation of confirmed immune-related disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Estimated to be from time of informed consent up to 5 years
  Overall survival will be determined as the time from the start of treatment with MEDI0562 until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune LLC, Study Director — MedImmune LLC
Locations (12):
- United States (11):
  - Research Site, La Jolla, California
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Research Site, Seoul, South Korea

REFERENCES:
- [Derived] Glisson BS, Leidner RS, Ferris RL, Powderly J, Rizvi NA, Keam B, Schneider R, Goel S, Ohr JP, Burton J, Zheng Y, Eck S, Gribbin M, Streicher K, Townsley DM, Patel SP. Safety and Clinical Activity of MEDI0562, a Humanized OX40 Agonist Monoclonal Antibody, in Adult Patients with Advanced Solid Tumors. Clin Cancer Res. 2020 Oct 15;26(20):5358-5367. doi: 10.1158/1078-0432.CCR-19-3070. Epub 2020 Aug 14. PMID 32816951